CLINICAL TRIAL: NCT04834245
Title: Evaluation of Diabetic Foot Wound Healing Using Hydrogel/Nano Silver-based Dressing vs. Traditional Dressing: A Prospective Randomized Control Study
Brief Title: Evaluation of Diabetic Foot Wound Healing Using Hydrogel/Nano Silver-based Dressing vs. Traditional Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Magda Bayoumi (Other)
Responsible Party: Sponsor-Investigator, Magda Bayoumi, Lecturer, Beni-Suef University
Organization: Beni-Suef University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: A12982019
Record Dates: First submitted 2021-04-01; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus
Keywords: Diabetic foot ulcer
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hydrogel/nano silver-based dressing (Experimental): hydrogel/nano silver-based dressing
  Interventions: Procedure: Hydrogel/nano silver-based dressing

INTERVENTIONS:
Procedure: Hydrogel/nano silver-based dressing — compare the effectiveness of using hydrogel/nano silver-based dressing vs. traditional dressing on diabetic foot wound healing.

SUMMARY:
Background: The wound dressings perform a crucial role in the cutaneous wounds' management due to their ability to protect wounds and promote dermal and epidermal tissue regeneration. Objective: the aim of the present study to evaluate the effectiveness of using hydrogel/nano silver-based dressing vs. traditional dressing on diabetic foot wound healing.

Approach: Sixty patients with type-2 diabetes hospitalized for diabetic foot wound treatment were recruited from selected Surgical departments at Kasr Al-Aini university hospital.

DETAILED DESCRIPTION:
Data Collection: The patients of group-I wounds were cleaned using normal saline; then, the wounds were closed firmly with hyderogel\nano silver dressing. The dressing was changed every two days according to dressing manufacture instruction. When the dressing was opened after three days, the wound was assessed for granulation tissue, wound, and discharge size.

The patients of group II wounds were dresses using a traditional method, cleaned by normal saline, use of betadine antiseptic; then they were secured with clean linen gauze. The dressing was changed once daily. The wound healing process of the two groups was then assessed for three consecutive weeks.

ELIGIBILITY:
Inclusion Criteria:

Diabetes Type I and Type II patient with diabetic foot ulcer age ranged 35-55 years old Willing to participate

Exclusion Criteria:

unwilling to participate.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
the percentage of a reduction rate of the diabetic foot ulcer after intervention | 3 Weeks
  assess of diabetic foot ulcers size "sq mm"

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No